CLINICAL TRIAL: NCT03975842
Title: Chronic Otitis Media With Effusion in Chronic Sinusitis With Polyps
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: 30138520
Record Dates: First submitted 2019-06-04; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyposis (CRSwNP)
Keywords: otitis media with effusion (OME); prevalence; risk factor; endoscopic nasal examination; otoscopic examination; pure-tone audiometry; tympanometry
MeSH Terms: conditions — Otitis Media with Effusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sinonasal and otologic evaluation — At onset, each participant had:
  * sinonasal evaluation (several nasal signs and symptoms were evaluated, bilateral endoscopic nasal examination, computed tomography (CT) of the sinuses when sinus surgery became necessary).
  * otologic evaluation (evaluation of middle ear status, documentations of personal history of otologic disease, otoscopic examination, pure-tone audiometry and tympanometry)

SUMMARY:
The relationship between otitis media with effusion (OME) and chronic rhinosinusitis with nasal polyposis (CRSwNP) remains unclear. A cross-sectional study of 80 consecutively presenting patients who were diagnosed with CRSwNP was conducted. The aim was to ascertain the prevalence of OME in CRSwNP patients, to determine whether the severity of CRSwNP affected OME, and to identify risk factors for OME in CRSwNP patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 15 years of age
* Presence of chronic rhinosinusitis with nasal polyposis (CRSwNP) previously diagnosed or diagnosed at study's onset by endoscopic nasal examination

Exclusion Criteria:

* Presence of a mucopurulent discharge or granuloma during endoscopic nasal examination

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic rhinosinusitis with nasal polyposis (CRSwNP)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The prevalence of OME in CRSwNP patients. | 2 years

IPD SHARING:
Plan to Share IPD: No